CLINICAL TRIAL: NCT02861287
Title: Economic Evaluation of the Use of Plerixafor for Autologous Hematopoietic Stem Cell Transplantation for Multiple Myeloma
Brief Title: Economic Evaluation of the Use of Plerixafor for Autologous HSC Transplantation for Multiple Myeloma
Acronym: PLERIXAFOR
Status: Completed | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: PLERIXAFOR-IPC 2013-002
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cost-Benefit Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study cohort: patients with Multiple Myeloma who underwent PBSC mobilization since December 2009 and who received plerixafor in line with inclusion criteria
  Interventions: Other: Economic evaluation
- Historical cohort: patients with Multiple Myeloma who underwent PBSC mobilization immediately prior to marketing authorization and clinical utilization of Plerixafor which is before December 2009 (over the 2007-2009 period)
  Interventions: Other: Economic evaluation

INTERVENTIONS:
Other: Economic evaluation

SUMMARY:
This study aims to realize an economic evaluation of the introduction of Plerixafor in addition to G-CSF and alternative options, in patients with multiple myeloma (MM) who failed or insufficiently mobilize peripheral blood stem and progenitor cells in response to G-CSF alone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with Multiple Myeloma who were eligible for high-dose melphalan supported with autologous hematopoietic stem cell transplantation (HSCT) as part of their treatment plan
* First mobilization attempt
* "rhG-CSF alone" mobilization regimen
* Failed mobilization as documented by an increase in CD34+ cell mobilization deemed insufficient to initiate apheresis (below 15/µL), after the 4 first injections of rhG-CSF that are administered in the evening

Exclusion Criteria:

* Age < 18 years;
* Primary diagnosis other than MM
* 2nd or subsequent mobilization attempt
* Patients who previously received HDCT + autologous HSCT
* Chemotherapy-based mobilization regimen
* Efficient mobilization, allowing for apheresis and collection of the target cell number (5x106 CD34+ cells/kg for every planned autologous transplantation as per institutional SOPs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will retrospectively review 60 electronic health records of patients who underwent peripheral blood stem cell mobilization for Multiple Myeloma, and who failed to achieve efficient and clinically meaningful mobilization in response to a well-conducted "G-CSF alone" regimen.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Cost-effectiveness analysis | 1 year
  The cost-effectiveness analysis will be performed using the collection of a transplantable graft as effectiveness criteria; the suitability of collected cell products for transplantation will be judged as per institutional criteria.
  Direct medical costs will be estimated by micro-costing, i.e. by measuring physical quantities (capital and labor) consumed for each patient and attributing corresponding monetary costs on the basis of average French prices. Costs (including room - inpatient and outpatient, drugs and laboratory tests) will be estimated on the basis of patients' medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Chabannon, MD PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli-Calmettes, Marseille, Bouches-du Rhône, France

IPD SHARING:
Plan to Share IPD: No